CLINICAL TRIAL: NCT03333122
Title: Prospective Evaluation of Patient Reported Outcomes and Satisfaction With Education in Breast Cancer Patients (PROS)
Brief Title: Assessment of Breast Cancer Patients Satisfaction and Health Related Quality of Life Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Dunya Atisha, MD, Henry Ford Health System
Other Study IDs: 11056
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Female
Keywords: Breast Cancer Breast-Q; Breast Reconstruction; Breast Conserving Therapy; Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Breast Conserving Therapy: Patient who undergo breast conserving therapy or breast conserving therapy with oncoplastic therapies will complete the BREAST-Q Lumpectomy survey module.
- Mastectomy: Patients who undergo mastectomy will complete the BREAST-Q Mastectomy survey module.
- Mastectomy with Reconstruction: Patient who undergo breast reconstruction will complete the BREAST-Q Reconstruction survey module. This group will be further subdivided based on implant or autologous tissue reconstruction.

SUMMARY:
The purpose of the study is to learn more about the quality of life and satisfaction with breast cancer surgical treatment and education from patient reported outcome data. The data and information obtained from breast cancer patients can be invaluable in counselling patients with a new diagnosis of breast cancer on their expected outcomes and results. The hypothesis is that using prospectively obtained data to guide surgical decision-making and optimize access to surgical procedures would improve the treatment of patients and would most likely positively impact the health-related quality of life in patients.

DETAILED DESCRIPTION:
This study will be a prospective observational study of women with newly diagnosed breast cancer. To date, there is little data in the literature assessing and comparing the outcomes associated with breast cancer surgical procedures. Information of satisfaction of patients with treatment, result, and breast cancer education they receive is particularly deficient. Therefore, breast cancer female patients will be recruited at Henry Ford Health System. Participants will voluntarily complete surveys electronically at specific points during their treatment and recovery process. Responses and satisfaction of quality of life will be collected and analyzed.

The BREAST-Q survey will be used to obtain patient reported outcomes.The surveys will be given preoperatively, at six months, one year, two years, and five years. Specific surveys will be given to the patients based on the treatment modality they receive.The groups are breast conserving therapy, mastectomy along, and mastectomy with reconstruction.The mastectomy with reconstruction group will be further subdivided based on implant or autologous tissue reconstruction. A survey adapted from the 'Patient Satisfaction with Cancer Treatment Education (PS-CaTE)' questionnaire will be administered at the preoperative and one year time point to evaluate satisfaction with their breast cancer education. PS-CaTE consists of two parts. Part one evaluates the patient's perception of the breast cancer education. Part two serves to elucidate the primary information sources the patients utilized by the patients. A demographic survey will also be given to patients preoperatively and postoperatively. Survey results will be analyzed to detect differences in health-related quality of life among the different treatments.

BREAST-Q surveys are health-related quality of life survey instruments developed to allow validated and reliable acquisition of patient reported outcomes.These surveys were meticulously crafted following internationally accepted guidelines as established by the Scientific Advisory Committee of the Medical Outcomes Trust and the U.S. Food and Drug Administration. The item list of this survey was developed from patient interviews, focus groups, expert panels, and literature review. Separate modules were developed for each treatment modality and include BREAST-Q Breast Conserving Therapy, BREAST-Q Mastectomy, BREAST-Q Reconstruction. These surveys have been used in major trials including the United Kingdom's National Health Service survey of 8,000 patients with mastectomy and mastectomy with reconstruction and FDA surveillance and longitudinal follow-up of patients with silicone breast implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients having surgery for breast cancer
* Treatment must be performed within the Henry Ford Health System
* Patients must be at least 18 years of age

Exclusion Criteria:

* Male gender
* Patients with non-operative management of breast cancer
* Patients who are unable to complete the surveys, either by choice or because of limited English, Spanish, or Arabic proficiency
* Patients who are unable to complete a preoperative survey
* Patients with Stage IV or metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of adult female patients who are diagnosed with breast cancer will be recruited from the Multidisciplinary Clinic at Henry Ford Health System.
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Compare health-related quality of life outcomes using condition specific surveys among women undergoing breast conserving therapy, mastectomy alone, or mastectomy with reconstruction | Up to 5 Years
  The BREAST-Q survey is used to determine differences in health-related of life between treatment groups.
Compare patient satisfaction with their treatment and result among women undergoing breast conserving therapy, mastectomy alone, or mastectomy with reconstruction | Up to 5 Years
  The BREAST-Q survey is used to detect differences in patient satisfaction among the groups.
Determine the effect of time on patient reported outcomes | Up to 5 Years
  Survey responses will be compared across time.
Patient satisfaction with breast cancer education and compare with source of information and socioeconomic status | Up to 1 Year
  PS-CaTE survey is administered to assess patient satisfaction with breast cancer education.

CONTACTS AND LOCATIONS:
Overall Officials: Dunya Atisha, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No